CLINICAL TRIAL: NCT03790514
Title: Alternative Therapy for Pain Management in Patients With Renal Colic: Heat Wrap
Brief Title: Heat Wrap for Renal Colic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Murat Gül, Assistant Professor, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AksarayUTRH
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Renal Colic
Keywords: Heat wrap
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Wrap Group (Experimental)
  Interventions: Other: Heat Wrap
- Control Group (Placebo Comparator)
  Interventions: Other: Heat Wrap

INTERVENTIONS:
Other: Heat Wrap — Commercially heat tapes ( without drugs) will be applied to patients.

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAIDs) (diclofenac, kotorolac, piroxicam) opioids (petidine, tramadol, fentanyl), paracetamol and topical agents (EMLA, diclofenal gel), have been shown to be effective in the treatment of renal colic . NSAIDs are commonly used to treat renal colic, but they can reduce renal blood flow and cause kidney damage. In addition, there are limitations in use in cases such as gastrointerstinal ulcers, hepatic insufficiency and chronic obstructive pulmonary disease. Gastrointestinal complications (ulcers, reflux, etc.) may cause hypersensitivity reactions (allergy) and coagulation disorders. On the other hand, opioids may cause nausea, vomiting, hypotension, sedation, dizziness and even respiratory depression. In addition to these pharmacological agents, stair-stroke, Turkish bath, blanket or hot water bag and local warming are now used in the treatment of renal colic in traditional methods.

Heat Wrap is an effective, natural solution designed to remove muscle pain with the help of heat and used regularly by physical therapists. The heat wrap is activated by air contact within a few minutes after its removal from its sheet and does not contain any drugs. It contains heat from the active iron particles in contact with air. After a few minutes of application, it begins to spread the natural, long-term (8 hours) heat by targeting the source of the pain. The patient satisfaction is high because it is odorless and thin.

In the literature, considering the success of heat therapy in patients with renal colic (bath entrance, electric blanket heating) in this study we have aimed to evaluate the efficacy of alternative treatment with pain-relieving alternative treatments with little potential for side effects and to see its applicability in daily treatment plans.

ELIGIBILITY:
Inclusion Criteria:

- Patients with renal colic

Exclusion Criteria:

* Pregnants
* Known allergies to heat tapes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Scale | 1 hour
  Self reported pain intensity (VAS 0-10) after applying heat wrap. Each item is scored between 0-10. While 0 shos no pain, 10 is the greatest pain the patient has experienced

CONTACTS AND LOCATIONS:
Locations (1):
- Murat Gül, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No